CLINICAL TRIAL: NCT06412107
Title: Somatic Acupressure on Fatigue-sleep Disturbance-depression Symptom Cluster in Breast Cancer Survivors: a Phase III Randomised Controlled Trial
Brief Title: Somatic Acupressure for Symptom Cluster Management in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Darwin University (Other)
Collaborators: Second Affiliated Hospital of Zunyi Medical University (Other); Zunyi Medical College (Other); University of Southern Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H22110; ETH2025-0294
Record Dates: First submitted 2024-02-26; First posted 2024-05-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasm Female; Symptom Cluster
Keywords: cancer; acupressure; fatigue; depression; insomnia
MeSH Terms: conditions — Syndrome; Neoplasms; Fatigue; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study can achieve a partial blind design for participants in the true and sham acupressure groups. Blind of outcome assessment will be also achieved in the true and sham intervention groups as all the questionnaires are patient-reported and the participants themselves will be the outcome assessors. Data analysis will be conducted by an independent statistician who are blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True acupressure group (Experimental): True self-acupressure plus routine methods of treatment and care.
  Interventions: Other: True acupressure; Other: Usual care
- Sham acupressure group (Sham Comparator): Same dose as the true acupressure group but on the sham acupoints plus routine methods of treatment and care.
  Interventions: Other: Sham acupressure; Other: Usual care
- Usual care group (Other): Routine methods of treatment and care.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: True acupressure — Participants will receive a 7-week true self-acupressure practice and a 12-week follow-up.
  Arms: True acupressure group
Other: Sham acupressure — Participants will receive a 7-week sham self-acupressure practice and a 12-week follow-up.
  Arms: Sham acupressure group
Other: Usual care — Routine methods of treatment and care along with an updated education booklet.

SUMMARY:
This study is designed following the updated Medical Research Council (MRC) Framework for Developing and Evaluating Complex Interventions. The goal of this randomized controlled trial (RCT) is to evaluate the effects, safety, and cost-effectiveness of an evidence-based somatic acupressure (SA) intervention on the fatigue-sleep disturbance-depression symptom cluster and quality of life among breast cancer survivors.

DETAILED DESCRIPTION:
Fatigue, sleep disturbance, and depression commonly co-occur in breast cancer (BC) survivors, forming a significant cluster known as the fatigue-sleep disturbance-depression symptom cluster (FSDSC). The FSDSC correlates notably with decreased everyday functioning and quality of life (QoL). Currently, there are no targeted pharmacological interventions available for alleviating the FSDSC in BC survivors. Additionally, concerns arise regarding the risks of drug-related adverse events and potential interactions with ongoing antineoplastic regimens when relying solely on pharmacological treatments. Consequently, nonpharmacological adjunct interventions have emerged as an alternative method. Somatic acupressure (SA) presents a promising nonpharmacological intervention for managing the FSDSC due to its advantages, including self-administration with minimal effort and time, lower cost, good tolerability, and minimal instruction required from clinical staff. However, the effectiveness of SA in improving the FSDSC in BC survivors remains uncertain. The proposed study follows the Medical Research Council (MRC) Framework for Developing and Evaluating Complex Intervention (the MRC Framework) to develop an evidence-based SA protocol to help with the better management of the FSDSC in BC survivors. The first phase identified and validated the most effective acupoint formula with the optimal SA duration and frequency based on multiple evidence bases. Subsequently, a well-designed phase II randomized controlled trial (RCT) was conducted. It demonstrated the feasibility of an evidence-based SA intervention protocol and its potentially positive effects on the FSDSC in BC survivors. The encouraging results, therefore, warrant further investigation through a large-scale RCT to ascertain the effects of SA on the FSDSC among BC survivors. The whole program is designed following the MRC Framework. Hence, the current study aims to evaluate the effects, safety, and cost-effectiveness of the SA protocol for managing the FSDSC in BC survivors through a phase III RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with early-stage female BC without distant metastases (from stage I to IIIa).
2. Have experienced at least moderate FSDSC with a score of ≥4 on an 0-10 point Numeric Rating Scale (0= 'no symptom',10= 'worst symptom') for fatigue, sleep disturbance and depression during the past month.
3. Had completed chemotherapy for at least one month and up to three years (to capture persistent symptoms)
4. Have no scheduled chemotherapy or radiotherapy during the study.
5. Be willing to participate in this study and consent in writing.

Exclusion Criteria:

1. Currently using pharmaceutical drugs (e.g., antidepressant medications or hypnotics) to treat symptoms of fatigue, sleep disturbance, or depression.
2. Inability (or difficulty) in following the study procedures and instructions due to being extremely weak and/or cognitively impaired.
3. Received any type of somatic acupressure interventions during the past six months.
4. Currently involved in any other studies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Fatigue | Baseline Assessments (T1); Immediately after completion of the 7-week intervention (T2); 12-week Follow-up (T3)
  The Brief Fatigue Inventory (BFI; 9 items) will be used to measure the participants' fatigue, with 0 = "no fatigue" and 10 = "fatigue as bad as you can imagine." The global score for the BFI is calculated as the mean value of these 9 items. A higher score indicates greater severity of fatigue.
Sleep disturbance | Baseline Assessments (T1); Immediately after completion of the 7-week intervention (T2); 12-week Follow-up (T3)
  The Pittsburgh Sleep Quality Index (PSQI; 19 items) will be used to assess sleep disturbance. A global (total) score is obtained from the sum of the seven component scores, with a possible range of 0 to 21 points. A higher total score indicates poorer sleep quality.
Depression | Baseline Assessments (T1); Immediately after completion of the 7-week intervention (T2); 12-week Follow-up (T3)
  The Hospital Anxiety and Depression Scale-Depression (HADS-D; 7 items; score range 0-21) will be used for evaluating depression. A higher score indicating greater severity of depression
Symptom cluster assessment: fatigue | Baseline Assessments (T1); Immediately after completion of the 7-week intervention (T2); 12-week Follow-up (T3)
  The 0-10 Numeric Rating Scale (0='no symptom', 10='worst symptom') will be used to assess fatigue.
Symptom cluster assessment: sleep disturbance | Baseline Assessments (T1); Immediately after completion of the 7-week intervention (T2); 12-week Follow-up (T3)
  The 0-10 Numeric Rating Scale (0='no symptom', 10='worst symptom') will be used to assess sleep disturbance.
Symptom cluster assessment: depression | Baseline Assessments (T1); Immediately after completion of the 7-week intervention (T2); 12-week Follow-up (T3)
  The 0-10 Numeric Rating Scale (0='no symptom', 10='worst symptom') will be used to assess depression.

SECONDARY OUTCOMES:
Patients' Quality of life | Baseline Assessments (T1); Immediately after completion of the 7-week intervention (T2); 12-week Follow-up (T3)
  The Functional Assessment of Cancer Therapy-Breast (FACT-B; 37 items) will be used for assessing the Patients' Quality of life. A summing-up of each FACT-B subscale creates the FACT-B total score, ranging from 0 to 148. A higher score indicates a better Quality of life.
Safety: adverse events | The adverse event will be assessed once it occurs during the study period, from the baseline to the end of 7 weeks.
  Adverse events will be collected through regular contact between the participant and the research assistant across the intervention period.
Economic evaluation | Weekly data collected across the 19 weeks.
  A within-trial economic evaluation will be conducted whereby clinical outcomes (fatigue-sleep disturbance-depression symptom cluster and quality of life) and cost data will be compared between the true intervention group and the usual care group over 19 weeks. Data on economic-related resource use will be captured using a bespoke questionnaire over 19 weeks from randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, PhD, Principal Investigator — University of Southern Queensland; Charles Darwin University
Locations (2):
- China (2):
  - The Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou

IPD SHARING:
Plan to Share IPD: No
As required by the Human Research Ethics Committee at the study sites, IPD will not be shared with other researchers. Only de-identified, aggregated group data will be used for the purposes of this study

REFERENCES:
- [Derived] Li M, Wang T, Liu XL, Deng RL, Kwok WH, Yao LQ, Tan JB. Somatic acupressure for the management of the fatigue-sleep disturbance-depression symptom cluster in breast cancer survivors: a study protocol for a phase III randomised controlled trial. BMJ Open. 2025 Mar 3;15(3):e089515. doi: 10.1136/bmjopen-2024-089515. PMID 40032405